CLINICAL TRIAL: NCT04717843
Title: Identification of New Markers of Atrial Myopathy in Patients With Embolic Stroke of Undetermined Source (ESUS) From MRI 4D Data
Acronym: IRM 4D-AVC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL20_0790
Record Dates: First submitted 2021-01-15; First posted 2021-01-22 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-06

CONDITIONS: Embolic Stroke of Undetermined Source
Keywords: Atrial Myopathy; Atrial Fibrillation; ESUS; MRI; blood velocity; left atrium
MeSH Terms: conditions — Atrial Fibrillation | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Patients with embolic strokes of undetermined source. (Experimental): Patients over 18 years old, with embolic strokes of undetermined source, fulfilling the TOAST criteria. The intervention consists of a 4D Flow MRI.
  Interventions: Other: 4D Flow MRI
- Patients with non-paroxysmal AF. (Experimental): Patients over 18 years old, with non-paroxysmal AF. The intervention consists of a 4D Flow MRI.
  Interventions: Other: 4D Flow MRI
- Heathy volunteers (Active Comparator): The control group will include volunteers over 45 years old with no history of cardio-vascular or neuro-vascular disease. The last will be certified by a pre inclusion protocol containing a medical consultation, a Holter ECG and a trans-thoracic echocardiography. The age of 45 was chosen to get comparable age group and set the analyses free of the age-related effect on the cardiac hemodynamic. The intervention consists of an ECG, holter ECG, Trans thoracic echocardiography ETT, Blood sample and 4D Flow MRI.
  Interventions: Other: 4D Flow MRI; Other: Medical consultation with 12 leads ECG; Other: Holter ECG; Other: Trans thoracic echocardiography; Biological: Blood sample
- ESUS and non-paroxysmal AF patients with cardiac MRI (Experimental): ESUS and non-paroxysmal AF patients (fulfilling the group 1 et 2 criteria) and who had had cardiac MRI, in a retrospective way. It corresponds to retrospective inclusion of patients which had MRI in the year before the beginning of the study.
  Interventions: Other: Standard MRI

INTERVENTIONS:
Other: 4D Flow MRI — Acquisitions of MR imagining with special contrast phase CMR sequences. There is no need for agent contrast injection. The CMR is performed at the time of inclusion.
  Arms: Heathy volunteers; Patients with embolic strokes of undetermined source.; Patients with non-paroxysmal AF.
Other: Medical consultation with 12 leads ECG — Collection of medical history, treatment, physical examination and realization of a 12 leads ECG.
  Arms: Heathy volunteers
Other: Holter ECG — 48 hours ECG recording
  Arms: Heathy volunteers
Other: Trans thoracic echocardiography — Trans thoracic echocardiography with standard measures performes in the core lab.
  Arms: Heathy volunteers
Biological: Blood sample — Blood sample in a peripheral vein, send to medical laboratory to dosage of NT pro BNP and troponin serum level.
  Arms: Heathy volunteers
Other: Standard MRI — Acquisitions of MR imagining
  Arms: ESUS and non-paroxysmal AF patients with cardiac MRI

SUMMARY:
Atrial myopathy is considered to be the underlying cause of a large proportion of embolic strokes of undetermined source. However, the definition of this atrial condition is not well delineated while its identification could lead to prescription on anticoagulation in order to avoid stroke recurences. This study aims to identify new markers of atrial myopathy and choosed a multi parametric approach with electrical, echographical, biological and 4D flow CMR derived markers.

ELIGIBILITY:
Inclusion Criteria:

Groupe1:Ischemic embolic stroke of undetermined source (ESUS) according to TOAST criteria (N =10)

* Age ≥ 18 years old
* Non-gap ischemic stroke diagnosed on MRI or CT scan of the brain (gap stroke defined as a cerebral infarction ≤ 1.5 cm / ≤2.0 cm on diffusion sequences).
* No major cardio-embolic source (episode of atrial fibrillation or flutter > 6min, intracardiac thrombus, LVEF <30 percent recent myocardial infarction (<4 weeks), mitral stenosis, valvular vegetation or infectious endocarditis).
* Absence of atherosclerosis causing stenosis ≥ 50 percent of the lumen of the intra or extra cranial arteries that vascularise the infarcted cerebral area.
* No other specific cause identified (arteritis, arterial dissection, migraine/vaso-spasm, toxic cause).
* Affiliation to a social security scheme
* Patient who signed the consent

Group 2: Non-paroxysmal AF (N=10)

* Age ≥ 18 years old
* Subject with documented non-paroxysmal AF
* Affiliation to a social security scheme
* Patient who signed the consent

Group 3: Healthy volunteers (N=10)

Pre-inclusion criteria :

* Age ≥ 45 years old
* Patient with no documented cardiac or neuro-vascular history
* Affiliation to a social security scheme
* Patient who signed the consent
* Registration on the VRB file (Volontaires Recherches Biomédicales, https://vrb.sante.gouv.fr) or response to the published announcement

Criteria for inclusion :

* ECG in sinus rhythm
* Holter ECG: no AF
* Normal Trans thoracic echocardiography
* Patient with no neuro-vascular history

Group 4: Stroke-ESUS or non-paroxysmal AF with cardiac MRI (N=10)

* Age ≥ 18 years old
* Subject with a documented stroke-ESUS or documented non-paroxysmal FA
* Subject with cardiac MRI
* Affiliation to a social security scheme
* Subject having given its non-opposition

Exclusion Criteria:

Groupe1: Ischemic embolic stroke of undetermined source (ESUS) according to TOAST criteria (N =10)

* Risk of pregnancy or pregnancy (proven on interrogation data or pregnancy test).
* Contraindication to MRI ferromagnetic material (in particular pacemaker, implantable defibrillator, cardiac valve prosthesis, cochlear implant, neuro-stimulator, implanted automated injection material, intraocular metallic foreign body, neurosurgical and vascular clips, claustrophobia)
* Less than 8 weeks after implantation of a stent
* Subject participating in another intervention research including a period of exclusion still in progress at the pre-inclusion stage.

Group 2: Non-paroxysmal AF (N=10)

* Risk of pregnancy or pregnancy (proven on interview data or pregnancy test).
* Contraindication to MRI ferromagnetic material (in particular pacemaker, implantable defibrillators, cardiac valve prosthesis, cochlear implant, neurostimulators, implanted automated injection equipment, intraocular metallic foreign body, neurosurgical and vascular clips, claustrophobia).
* Less than 8 weeks after implantation of a stent
* Subject participating in another intervention research including a period of exclusion still in progress at the pre-inclusion stage.

Group 4: Stroke-ESUS or non paroxysmal AF with cardiac MRI (N=10)

* History of neuro-vascular or cardiac pathology
* Risk of pregnancy or pregnancy (proven on interrogation data or pregnancy test).
* Contraindication to MRI (ferromagnetic material (in particular pacemaker, implantable defibrillator, cardiac valve prosthesis, cochlear implant, neuro-stimulator, implanted automated injection material, intraocular metallic foreign body, neurosurgical and vascular clips, claustrophobia)
* Subject participating in another intervention research including a period of exclusion still in progress at the pre-inclusion stage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Mean flow velocities in the left atrium | One Day
  Velocity magnitude (cm/s) for all atrial voxels and all cardiac frames will be plotted in a histogram and normalized by the total number of voxels to allow comparisons between subjects

SECONDARY OUTCOMES:
Maximal flow velocities in the left atrium | One Day
  Velocity magnitude (cm/s) for all atrial voxels and all cardiac frames will be plotted in a histogram and normalized by the total number of voxels to allow comparisons between subjects. Local peak velocity will be obtained by averaging 5 percent of all maximum values.
Left atrium stasis | One Day
  Velocity magnitude (cm/s) for all atrial voxels and all cardiac frames will be plotted in a histogram and normalized by the total number of voxels to allow comparisons between subjects. Local peak velocity will be obtained by averaging 5 percent of all maximum values
Vortex size | One Day
  Vortices in the isolated LA chamber were detectedusing the Lambda2 (λ2) method, which is an objective and widelyaccepted method to identify 3D vortice.
Left atrium volume | One Day
  Extracted from 3D MR reconstruction, expressed in mL/m2 of body surface area.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe CHEVALIER, Pr, Principal Investigator — Chief of the Arrhythmia Unit at the Academic Hospital of Lyon
Locations (3):
- France (3):
  - Service d'urgences neuro-vasculaires, service de neurologie vasculaire Hôpital neurologique Pierre Wertheimer, Bron
  - Service Imagerie médicale Hôpital neurologique Pierre Wertheimer, Bron
  - Service rythmologie, Hôpital cardiologique Louis Pradel, Bron